CLINICAL TRIAL: NCT00005751
Title: Endothelial Vasomotor Function in the Framingham Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5081; R01HL060040 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine whether the presence of endothelial dysfunction is an independent risk factor for cardiovascular disease events.

DETAILED DESCRIPTION:
BACKGROUND:

Current research suggests that loss of the vasodilator, anti-thrombotic, and anti-inflammatory properties of the vascular endothelium plays a dynamic role in the pathogenesis of cardiovascular disease. Impaired endothelial function, including impaired nitric oxide-dependent vasodilation is associated with cardiovascular disease risk factors. Further, there is growing evidence that endothelial function can be improved by risk modification. However, the available studies have not definitively resolved the issue of the cross-sectional correlates of endothelial dysfunction because they have been limited to small samples of highly selected patients. For example, it remains unclear whether hypercholesterolemia, hypertension, or elevated glucose levels are independent determinants of endothelial dysfunction. Most importantly, no study has shown a relation between endothelial dysfunction and increased cardiovascular risk. Such a demonstration would increase our understanding of the pathogenesis of cardiovascular disease and aid clinicians in identifying high risk individuals who would benefit most from intervention.

DESIGN NARRATIVE:

Using non-invasive brachial artery ultrasound, endothelial function was examined in about 3,800 men and women of the Framingham Heart Study. The cross-sectional correlates of endothelial function with known coronary risk factors were examined and cross-sectional analyses were performed on the relation of endothelial function to prevalent cardiovascular disease. Observations were made of the adjusted relation of endothelial function to incident and recurrent cardiovascular events. The central hypothesis was that the presence of endothelial dysfunction was an independent risk factor for cardiovascular disease events.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-12; Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Benjamin — Boston University

REFERENCES:
- [Background] Vita JA, Keaney JF Jr. Endothelial function: a barometer for cardiovascular risk? Circulation. 2002 Aug 6;106(6):640-2. doi: 10.1161/01.cir.0000028581.07992.56. No abstract available. PMID 12163419
- [Background] Benjamin EJ, Larson MG, Keyes MJ, Mitchell GF, Vasan RS, Keaney JF Jr, Lehman BT, Fan S, Osypiuk E, Vita JA. Clinical correlates and heritability of flow-mediated dilation in the community: the Framingham Heart Study. Circulation. 2004 Feb 10;109(5):613-9. doi: 10.1161/01.CIR.0000112565.60887.1E. PMID 14769683